CLINICAL TRIAL: NCT06195852
Title: Maximizing the Reach of Universal Child Sexual Abuse Prevention: An Equivalence Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low participation rates from school entities invited to participate in research.
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21HD110822 (NIH)
Record Dates: First submitted 2023-12-08; First posted 2024-01-08 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Child Sexual Abuse
Keywords: prevention; universal prevention; school-based intervention; Safe Touches

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Safe Touches (Active Comparator): Delivered by 2 facilitators in a classroom by utilizing live puppet skits
  Interventions: Behavioral: Usual Safe Touches
- Modified Safe Touches (Experimental): Delivered by 1 facilitator in the classroom by utilizing prerecorded workshop skit videos
  Interventions: Behavioral: Modified Safe Touches

INTERVENTIONS:
Behavioral: Usual Safe Touches — The in-person Safe Touches workshop is delivered in the classroom by 2 facilitators with live puppet skits, as designed.
  Arms: Usual Safe Touches
Behavioral: Modified Safe Touches — The modified Safe Touches workshop will be delivered by 1 facilitator in the classroom by utilizing prerecorded workshop skit videos.
  Arms: Modified Safe Touches

SUMMARY:
The goal of this clinical trial is to test the equivalence of two delivery modalities of a universal child sexual abuse prevention program, Safe Touches: usual vs. modified. The aims are to:

1. Determine the equivalence of effectiveness between usual and modified Safe Touches
2. Assess the maintenance of gains between usual and modified Safe Touches
3. Examine factors that may impact the future dissemination and implementation

DETAILED DESCRIPTION:
Child sexual abuse (CSA) is a public health problem affecting 1 in 5 girls and 1 in 12 boys before age 18. National estimates indicate children ages 7 to 13 are at highest risk for CSA and CSA is associated with lifelong negative sequelae. School-based prevention programs offer cost-effective universal programming teaching students an array of personal safety skills. Several programs have demonstrated effectiveness in increasing children's knowledge of self-protection, and some have been linked with facilitating disclosures, including Safe Touches. Effectiveness notwithstanding, the programmatic reach of universal school-based programs is limited by the inherent reliance on school infrastructure and a dearth of available alternative delivery modalities. The current study is designed to address this gap by leveraging an existing partnership between university-based researchers (NYU), the Safe Touches model developer (NYSPCC), and community-based organizations with active implementations of Safe Touches. The study will use a rigorous cluster randomized design to determine the equivalence of effectiveness between two delivery modalities of Safe Touches: as usual vs. modified. The usual workshop will be delivered by two facilitators with live puppet skits, as designed (N=90). Whereas, the modified workshop will be delivered by one facilitator utilizing pre recorded skit videos (N=90). The research team will determine the equivalence of concept learning acquisition (Aim 1) and retention (Aim 2) among students in classrooms that receive the as usual or modified workshop. To conclude equivalence, it is important to examine factors that may impact future dissemination and implementation, specifically program adoption among school personnel and implementation fidelity (Aim 3). Study findings will inform the ongoing development of effective CSA prevention programs and policy decisions regarding the sustainable integration of such programs within schools. Given the scope and burden of CSA, especially among elementary aged students, it is a public health priority to efficiently disseminate effective school-based prevention programs on a wide scale.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in a second grade classroom participating in the research
* Native English speaker
* Parental permission to participate in the research

Exclusion Criteria:

* Not enrolled in a second grade classroom participating in the research
* Non-native English speaker
* No parental permission to participate in the research

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
Modified Children's Knowledge of Abuse Questionnaire | Pre-workshop, immediately post-workshop, 1-month follow up
  6-items rated on 3- point scale (Yes, Unsure, No) where higher scores indicate a greater knowledge of safe and unsafe touches

CONTACTS AND LOCATIONS:
Overall Officials: Kate Guastaferro, PhD, MPH, Principal Investigator — New York University
Locations (4):
- United States (4):
  - Weller Health Education at Lehigh Valley Health Network, Allentown, Pennsylvania
  - Northern Dauphin County YMCA, Elizabethville, Pennsylvania
  - Centre County (Centre Safe & Youth Service Bureau), State College, Pennsylvania
  - York County Children's Advocacy Center, York, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guastaferro K, Melchior MS, Heng S, Trudeau J, Holloway JL. Maximizing the reach of universal child sexual abuse prevention: Protocol for an equivalence trial. Contemp Clin Trials Commun. 2024 Jul 31;41:101345. doi: 10.1016/j.conctc.2024.101345. eCollection 2024 Oct. PMID 39188413